CLINICAL TRIAL: NCT03609190
Title: Brain Activation Patterns Under Emotional and Neurochemic Stimulation With Ketamine: A Multimodal Neuroimaging Study
Brief Title: A Multimodal Neuroimaging Study of Brain Activation Patterns Under Ketamine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Milan Scheidegger, Principal Investigator, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E-31/2008
Record Dates: First submitted 2018-07-13; First posted 2018-08-01 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): i.v. infusion of 0.25 mg/kg S-ketamine over 40 min
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): i.v. infusion of NaCl over 40 min
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — i.v. infusion of 0.25 mg/kg S-ketamine over 40 min
  Arms: Ketamine
Drug: Placebo — i.v. infusion of NaCl over 40 min
  Arms: Placebo

SUMMARY:
The aim of the project is to establish a multimodal imaging approach for the investigation of the neural mechanisms underlying neuroreceptor regulation, glutamatergic metabolism and brain function that are of particular relevance for major depressive disorder (MDD) and that can be translated into clinical applications.

There is growing evidence for imbalance with regard to glutamatergic neurotransmission in stress-related affective disorders. Further support for the hypothesis that dysfunctional glutamatergic signaling underlies major depressive disorder, and indeed that its reversal constitutes a potential efficacious mechanism of action, is provided by the evidence that pharmacological compounds active at the N-methyl-D-aspartate (NMDA) ionotropic glutamate receptor such as ketamine exert rapid antidepressant effects. As a tool compound ketamine enables the safe investigation of the brain region-specific effects of NMDA receptor antagonism in terms of glutamatergic neurotransmission, brain function and the association of these neural changes with emotional state, thereby allowing for increased understanding of the therapeutic mechanism of action.

The possibility to simultaneously study brain perfusion (arterial spin labeling), functional brain activity (fMRI) and connectivity (resting state fMRI), neurometabolism (proton magnetic resonance spectroscopy) and metabotropic glutamate receptor densities (positron emission tomography) will unravel their functional interplay in the mechanisms underlying the regulation of mood and cognition. Combining those imaging modalities with treatment interventions in healthy subjects and depressed patients, this project aims at providing insight into the neuropharmacological effects of ketamine and its antidepressant properties.

ELIGIBILITY:
Inclusion Criteria:

* treatment resistant depressive episode
* no restrictions regarding antidepressant medication

Exclusion Criteria:

* lifetime antidepressant treatment with ketamine
* lifetime recreational use of ketamine
* cardiovascular diseases such as hypertonia, cardiac insufficiency or myocardial infarct in the past six months
* insufficiently treated anemia
* hyper- or hypothyroidism
* lifetime increased intracranial pressure or glaucoma
* chronic physical diseases
* hepatorenal dysfunction
* any relevant psychiatric or neurological comorbidity, in particular dementia, epileptic seizures (lifetime), schizophrenia (lifetime), psychosis (lifetime), or post-traumatic stress disorder (current).
* acute suicidality
* substance abuse disorders
* recent heart or head surgery
* metallic body implants
* agoraphobia
* pregnancy
* left handedness

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in functional reactivity to emotional stimuli | Change from baseline to 24h-post infusion
  fMRI BOLD
Change in glutamate concentrations in prefrontal cortex | Change from baseline to 24h-post infusion
  1H-MRS
Change in resting-state functional connectivity | Change from baseline to 24h-post infusion
  rsfMRI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herrera-Melendez A, Stippl A, Aust S, Scheidegger M, Seifritz E, Heuser-Collier I, Otte C, Bajbouj M, Grimm S, Gartner M. Gray matter volume of rostral anterior cingulate cortex predicts rapid antidepressant response to ketamine. Eur Neuropsychopharmacol. 2021 Feb;43:63-70. doi: 10.1016/j.euroneuro.2020.11.017. Epub 2020 Dec 11. PMID 33309459
- [Derived] Gartner M, Aust S, Bajbouj M, Fan Y, Wingenfeld K, Otte C, Heuser-Collier I, Boker H, Hattenschwiler J, Seifritz E, Grimm S, Scheidegger M. Functional connectivity between prefrontal cortex and subgenual cingulate predicts antidepressant effects of ketamine. Eur Neuropsychopharmacol. 2019 Apr;29(4):501-508. doi: 10.1016/j.euroneuro.2019.02.008. Epub 2019 Feb 26. PMID 30819549